CLINICAL TRIAL: NCT01770353
Title: A Phase I Study in Patients Treated With MM-398 (Nanoliposomal Irinotecan, Nal-IRI) to Determine Tumor Drug Levels and to Evaluate the Feasibility of Ferumoxytol Magnetic Resonance Imaging to Measure Tumor Associated Macrophages and to Predict Patient Response to Treatment
Brief Title: MM-398 (Nanoliposomal Irinotecan, Nal-IRI) to Determine Tumor Drug Levels and to Evaluate the Feasibility of Ferumoxytol Magnetic Resonance Imaging to Measure Tumor Associated Macrophages and to Predict Patient Response to Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MM-398-01-01-02
Record Dates: First submitted 2012-12-19; First posted 2013-01-17 (Estimated); Results first posted 2019-10-28 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Solid Tumors; ER/PR Positive Breast Cancer; Triple Negative Breast Cancer; Metastatic Breast Cancer With Active Brain Metastasis
Keywords: solid tumors; Triple Negative Breast Cancer; Colorectal Cancer; MM-398; nanoliposomal irinotecan; Ferumoxytol; ER/PR positive Breast Cancer; Pancreatic Cancer; Ovarian Cancer; Gastric Cancer; Gastro-Esophageal Junction Adenocarcinoma; Head and Neck Cancer; TNBC
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Colorectal Neoplasms; Pancreatic Neoplasms; Ovarian Neoplasms; Stomach Neoplasms; Head and Neck Neoplasms | interventions — Ferrosoferric Oxide; irinotecan sucrosofate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- Pilot Phase: Ferumoxytol followed by MM-398 (Experimental): Ferumoxytol 5 mg/kg IV at the rate of 1 mL/sec, given once on Day 1. MM-398 IV over 90 min on Days 1 and 15 of every 4 week cycle
  Interventions: Drug: Ferumoxytol; Drug: MM-398
- Expansion Phase: Ferumoxytol followed by MM-398 (Experimental): Ferumoxytol 5 mg/kg IV at the rate of 1 mL/sec, given once on Day 1. MM-398 IV over 90 min dose 1 on Days 1 and 15 of every 4 week cycle Cohort 1: ER and/or PR-positive BC Cohort 2: TNBC Cohort 3: BC with active brain metastasis
  Interventions: Drug: Ferumoxytol; Drug: MM-398

INTERVENTIONS:
Drug: Ferumoxytol — Ferumoxytol 5 mg/kg IV as a single bolus injection, given once.
Drug: MM-398 — MM-398 IV over 90 min every 2 weeks, until progressive disease or intolerable toxicity

SUMMARY:
This is a Phase I study to understand the biodistribution of MM-398 and to determine the feasibility of using Ferumoxytol as a tumor imaging agent.

DETAILED DESCRIPTION:
This study is conducted over two phases.

Pilot Phase: This study will enroll approximately 12 patients, up to 20 in total in the Pilot Phase and 30 patients in the Expansion Phase. The first three patients that are enrolled in the Pilot Phase can have any solid tumor type; however subsequent patients must have Non-small cell lung cancer (NSCLC), Colorectal cancer (CRC), Triple negative breast cancer (TNBC), Estrogen Receptor/Progesterone Receptor (ER/PR) positive breast cancer, pancreatic cancer, ovarian cancer, gastric cancer, gastro-oesophageal junction adenocarcinoma or head and neck cancer. No more than three patients with ER/PR positive breast cancer can be enrolled in the Pilot Phase and similar restrictions may be placed on other tumor types to ensure a heterogeneous population.

Expansion Phase: The expansion will enroll patients with advanced metastatic breast cancer into three cohorts of 10 patients each depending on sub-type of breast cancer:

Cohort 1: ER and/or PR-positive breast cancer Cohort 2: TNBC Cohort 3: BC with active brain metastasis

ELIGIBILITY:
Inclusion Criteria:

All subjects:

* Pathologically confirmed diagnosis of solid tumors
* Metastatic disease
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 1
* Adequate bone marrow, hepatic and renal function
* Normal Electrocardiogram (ECG)
* 18 years of age or above
* Able to understand and sign informed consent

Pilot study only:

- CRC, TNBC, ER/PR Breast Cancer, NSCLC, Pancreatic Cancer, Ovarian Cancer, Gastric Cancer, Gastroesophageal Junction (GEJ) adenocarcinoma, Head and Neck Cancer

Expansion Phase Additional Criteria:

* Locally advanced or metastatic breast cancer
* Received at least one cytotoxic therapy in the locally advanced and metastatic setting
* Received ≤ 5 prior lines of chemotherapy in the metastatic setting
* Candidate for chemotherapy

Expansion Phase Cohort 3 additional inclusion criteria:

* Breast cancer with active brain metastasis
* Neurologically stable

Exclusion Criteria:

* Active Central nervous system (CNS) metastasis (applies to pilot phase and expansion phase cohort 1 and 2 only)
* Clinically significant GI disorders
* Prior irinotecan or bevacizumab therapy within last 6 months and for Expansion Phase patients, have received any prior treatment with Topol inhibitor
* Known hypersensitivity to MM-398 or ferumoxytol
* Inability to undergo MRI
* Active infection
* Pregnant or breast feeding
* Prior chemotherapy administered within 3 weeks, or within a time interval less than at least 5 half-lives of the agent, whichever is longer, prior to the first scheduled day of dosing in this study
* Received radiation therapy in the last 14 days
* Treated with parenteral iron in the previous 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-11; Primary Completion 2018-10-02 (Actual); Study Completion 2018-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (7):
- United States (7):
  - Mayo Clinic, Scottsdale, Arizona
  - HonorHealth, Scottsdale, Arizona
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Moffitt Cancer Center, Tampa, Florida
  - University of Michighan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - UNC- Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina

REFERENCES:
- [Derived] Ravi H, Arias-Lorza AM, Costello JR, Han HS, Jeong DK, Klinz SG, Sachdev JC, Korn RL, Raghunand N. Pretherapy Ferumoxytol-enhanced MRI to Predict Response to Liposomal Irinotecan in Metastatic Breast Cancer. Radiol Imaging Cancer. 2023 Mar;5(2):e220022. doi: 10.1148/rycan.220022. PMID 36734848
- [Derived] Sachdev JC, Munster P, Northfelt DW, Han HS, Ma C, Maxwell F, Wang T, Belanger B, Zhang B, Moore Y, Thiagalingam A, Anders C. Phase I study of liposomal irinotecan in patients with metastatic breast cancer: findings from the expansion phase. Breast Cancer Res Treat. 2021 Feb;185(3):759-771. doi: 10.1007/s10549-020-05995-7. Epub 2020 Nov 17. PMID 33201358

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Six study centres in the United States recruited subjects into this Phase 1, 2-phase, non-comparative, open-label study. Each phase consisted of 4 stages: screening, ferumoxytol (FMX) treatment, irinotecan liposome injection (MM-398) treatment and follow-up (30 days after last dose).
Pre-assignment Details: Subjects with solid tumours were recruited to the Pilot phase. Subjects with locally advanced or metastatic breast cancer (BC) were recruited to the Expansion phase which consisted of 3 cohorts dependent on BC tumour sub-types and the presence of active brain metastases. Data was combined into 1 arm for the Expansion Phase as all subjects had BC.
Groups:
- Pilot Phase: FMX Then MM-398: FMX phase: Subjects received a single bolus intravenous (IV) injection of 5 milligrams per kilogram (mg/kg) FMX (up to 510 mg) on Day 1. Subjects underwent FMX magnetic resonance imaging (MRI) scans and pre-MM-398 treatment biopsies on Days 1 to 4.
  MM-398 Treatment phase: Within 7 days of the FMX infusion, subjects received up to 70 milligrams per square metre (mg/m^2) MM-398 free base equivalent (FBE) (Cycle 1 Day 1 [C1D1]) administered as an IV infusion over 90 minutes, repeated every 2 weeks until disease progression, unacceptable toxicity or withdrawal of consent.
- Expansion Phase: FMX Then MM-398: FMX phase: Subjects received an IV infusion of 5 mg/kg FMX (up to 510 mg) administered over a minimum of 15 minutes on Day 1. Subjects underwent FMX-MRI scans and a pre-MM-398 treatment biopsy on Days 1 to 2.
  MM-398 Treatment phase: Within 7 days of the FMX infusion, subjects received up to 70 mg/m^2 MM-398 FBE (C1D1) administered as an IV infusion over 90 minutes, repeated every 2 weeks until disease progression, unacceptable toxicity or withdrawal of consent.
  Cohort 1: Oestrogen receptor (ER) and/or progesterone receptor (PR)-positive BC and human epidermal growth factor receptor 2 (HER-2) negative BC.
  Cohort 2: Triple negative BC (TNBC). Cohort 3: BC with active brain metastasis.
Period: Overall Study
Arm/Group | Pilot Phase: FMX Then MM-398 | Expansion Phase: FMX Then MM-398
Started | 15 | 30
Received FMX (2 subjects in Pilot + 1 in Expansion died due to progressive disease before MM-398 treatment) | 15 (2 subjects excluded from MM-398 safety population.) | 30 (1 subject excluded from MM-398 safety population.)
Received FMX and MM-398 (MM-398 safety population.) | 13 | 29
Completed (Received MM-398 treatment up to disease progression.) | 9 | 18
Not Completed | 6 | 12
Not completed — Progressive disease | 2 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Physician Decision | 0 | 3
Not completed — Clinical deterioration | 3 | 6
Not completed — Toxicity related diarrhoea + progression | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for the safety population which included all subjects who received at least 1 dose of FMX or MM-398.
Groups:
- Pilot Phase: FMX Then MM-398: FMX phase: Subjects received a single bolus IV injection of 5 mg/kg FMX (up to 510 mg) on Day 1. Subjects underwent FMX-MRI scans and pre-MM-398 treatment biopsies on Days 1 to 4.
  MM-398 Treatment phase: Within 7 days of the FMX infusion, subjects received up to 70 mg/m^2 MM-398 FBE (C1D1) administered as an IV infusion over 90 minutes, repeated every 2 weeks until disease progression, unacceptable toxicity or withdrawal of consent.
- Expansion Phase: FMX Then MM-398: FMX phase: Subjects received an IV infusion of 5 mg/kg FMX (up to 510 mg) administered over a minimum of 15 minutes on Day 1. Subjects underwent FMX-MRI scans and a pre-MM-398 treatment biopsy on Days 1 to 2.
  MM-398 Treatment phase: Within 7 days of the FMX infusion, subjects received up to 70 mg/m^2 MM-398 FBE (C1D1) administered as an IV infusion over 90 minutes, repeated every 2 weeks until disease progression, unacceptable toxicity or withdrawal of consent.
  Cohort 1: ER and/or PR-positive BC and HER-2 negative BC. Cohort 2: TNBC. Cohort 3: BC with active brain metastasis.
- Total: Total of all reporting groups
Arm/Group | Pilot Phase: FMX Then MM-398 | Expansion Phase: FMX Then MM-398 | Total
Number analyzed (Participants) | 15 | 30 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 25 | 34
  >=65 years | 6 | 5 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 30 | 41
  Male | 4 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 13 | 27 | 40
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 2 | 2
  White | 14 | 23 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Pilot Phase: Tumour Levels of Irinotecan and SN-38 at Cycle 1 Day 4
Description: Two tumour biopsies were collected 72 hours after the first MM-398 IV infusion during Cycle 1 of the MM-398 Treatment phase of the Pilot phase for determination of tumour levels of irinotecan and SN-38 (an active metabolite). The lesions selected for biopsy were based on the results of the FMX-MRI obtained on Days 1, 2 and 4 of the FMX phase, and were collected from a previously non-biopsied lesion. The first core biopsy was taken in the region of the tumour that showed the greatest signal change on either the T2 or T1 sequences, based on FMX-MRI. The second core biopsy was taken from the region that showed the least signal change based on FMX-MRI, avoiding areas of necrosis.
Time Frame: At Cycle 1 Day 4 in the Pilot phase.
Population: The efficacy evaluable population included all subjects who received at least 1 dose of MM-398.
Measure: Mean (Standard Deviation); unit: nanograms per gram (ng/g)
Arm/Group | Pilot Phase: FMX Then MM-398
Number analyzed (Participants) | 13
nanograms per gram (ng/g)
  Irinotecan | 4253 (3600)
  SN-38 | 38.1 (91.5)

2. Primary Outcome: Expansion Phase: Impact of the Quality of MRI Scan on Tumour Evaluation
Description: Feasibility of FMX quantitation in tumour lesion was assessed through the acquisition of baseline (pre-FMX dose) and follow-up (post FMX dose) scans of sufficient quality to enable quantitative analysis to be performed. Quality was assessed by summarising scans as adequate for tumour evaluation or suboptimal but for which evaluation was completed for evaluation. Two FMX-MRI scans were taken on Day 1 (pre-FMX dosing) and on Day 2 (16-24 hours post dose) of the FMX phase. One MRI scan was also taken at 1-4 hours post FMX dose (Day 1 of FMX phase) and at 2 weeks post FMX dose (Day 15 of the MM-398 phase). It was possible for a subject to have 2 FMX-MRI scans for the same visit and timepoint corresponding to a scan target location. The number of MRI scan results that were assessed to be adequate or suboptimal at each timepoint are presented.
Time Frame: Expansion phase Cycle 1: Pre FMX dose, 1-4 hours post FMX dose, 16-24 hours post FMX dose, 2 weeks Post FMX dose.
Population: The pharmacodynamic evaluable population included all subjects who received at least 1 dose of MM-398 and who had pre-treatment FMX-MRI scan(s) and radiological scans at 8 weeks.
Measure: Number; unit: examined scans
Units Other Than Participants: Scans
Groups:
- Expansion Phase: Cohort 1: Subjects with ER and/or PR-positive BC and HER-2 negative BC.
  FMX phase: Subjects received an IV infusion of 5 mg/kg FMX (up to 510 mg) administered over a minimum of 15 minutes on Day 1. Subjects underwent FMX-MRI scans and a pre-MM-398 treatment biopsy on Days 1 to 2.
  MM-398 Treatment phase: Within 7 days of the FMX infusion, subjects received up to 70 mg/m^2 MM-398 FBE (C1D1) administered as an IV infusion over 90 minutes, repeated every 2 weeks until disease progression, unacceptable toxicity or withdrawal of consent.
- Expansion Phase: Cohort 2: Subjects with TNBC.
  FMX phase: Subjects received an IV infusion of 5 mg/kg FMX (up to 510 mg) administered over a minimum of 15 minutes on Day 1. Subjects underwent FMX-MRI scans and a pre-MM-398 treatment biopsy on Days 1 to 2.
  MM-398 Treatment phase: Within 7 days of the FMX infusion, subjects received up to 70 mg/m^2 MM-398 FBE (C1D1) administered as an IV infusion over 90 minutes, repeated every 2 weeks until disease progression, unacceptable toxicity or withdrawal of consent.
- Expansion Phase: Cohort 3: Subjects with BC with active brain metastasis.
  FMX phase: Subjects received an IV infusion of 5 mg/kg FMX (up to 510 mg) administered over a minimum of 15 minutes on Day 1. Subjects underwent FMX-MRI scans and a pre-MM-398 treatment biopsy on Days 1 to 2.
  MM-398 Treatment phase: Within 7 days of the FMX infusion, subjects received up to 70 mg/m^2 MM-398 FBE (C1D1) administered as an IV infusion over 90 minutes, repeated every 2 weeks until disease progression, unacceptable toxicity or withdrawal of consent.
Arm/Group | Expansion Phase: Cohort 1 | Expansion Phase: Cohort 2 | Expansion Phase: Cohort 3
Number analyzed (Participants) | 7 | 5 | 6
Number analyzed (Scans) | 7 | 5 | 11
examined scans
  Pre-FMX Dose (1): adequate | 4 | 3 | 7
  Pre-FMX Dose (1): suboptimal | 3 | 2 | 4
  Pre-FMX Dose (2): adequate: number analyzed (Scans) | 1 | 2 | 0
  Pre-FMX Dose (2): adequate | 0 | 1 |
  Pre-FMX Dose (2): suboptimal: number analyzed (Scans) | 1 | 2 | 0
  Pre-FMX Dose (2): suboptimal | 1 | 1 |
  1-4 hours Post FMX: adequate: number analyzed (Scans) | 6 | 2 | 7
  1-4 hours Post FMX: adequate | 4 | 1 | 5
  1-4 hours Post FMX: suboptimal: number analyzed (Scans) | 6 | 2 | 7
  1-4 hours Post FMX: suboptimal | 2 | 1 | 2
  16-24 hours Post FMX (1): adequate: number analyzed (Scans) | 7 | 5 | 10
  16-24 hours Post FMX (1): adequate | 4 | 3 | 6
  16-24 hours Post FMX (1): suboptimal: number analyzed (Scans) | 7 | 5 | 10
  16-24 hours Post FMX (1): suboptimal | 3 | 2 | 4
  16-24 hours Post FMX (2): adequate: number analyzed (Scans) | 1 | 0 | 0
  16-24 hours Post FMX (2): adequate | 0 |  |
  16-24 hours Post FMX (2): suboptimal: number analyzed (Scans) | 1 | 0 | 0
  16-24 hours Post FMX (2): suboptimal | 1 |  |
  Post FMX Day 15: adequate: number analyzed (Scans) | 1 | 3 | 0
  Post FMX Day 15: adequate | 0 | 2 |
  Post FMX Day 15: suboptimal: number analyzed (Scans) | 1 | 3 | 0
  Post FMX Day 15: suboptimal | 1 | 1 |

3. Primary Outcome: Expansion Phase: Best Overall Tumour Response (BOR) by Tumour FMX Uptake Classification at 16 - 24 Hours Post-FMX Dose
Description: FMX tumour uptake was classified as 'low tumour uptake' or 'high tumour uptake', and was determined for 16 to 24-hours post-FMX dosing. The FMX uptake in a subject's lesions was classified using the median of the baseline-corrected FMX values at that timepoint across all subjects. The best radiological overall tumour response to MM-398 from the beginning to the end of the study was assessed using both the Investigator and imaging results per Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1 (Non-central nervous system [CNS] assessments; Cohorts 1, 2 and 3). Tumour response was classified as a Complete Response (CR), Partial Response (PR), Stable Disease (SD) or Progressive Disease (PD). BOR is presented by tumour uptake classification at 16-24 hours post-FMX dose by cohort for the non-CNS RECIST assessment.
Time Frame: Expansion phase: C1D2 FMX phase, and every 8 weeks for RECIST assessments from C1D1 until disease progression, unacceptable toxicity or withdrawal of consent.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Expansion Phase: Cohort 1 | Expansion Phase: Cohort 2 | Expansion Phase: Cohort 3
Number analyzed (Participants) | 7 | 5 | 6
Participants
  High tumour uptake and CR | 1 | 0 | 0
  High tumour uptake and PR | 1 | 3 | 0
  High tumour uptake and SD | 0 | 2 | 0
  High tumour uptake and Non-CR/Non-PD | 0 | 0 | 0
  High tumour uptake and PD | 2 | 0 | 0
  Low tumour uptake and CR | 1 | 0 | 1
  Low tumour uptake and PR | 1 | 0 | 2
  Low tumour uptake and SD | 1 | 0 | 2
  Low tumour uptake and Non-CR/Non-PD | 0 | 0 | 0
  Low tumour uptake and PD | 0 | 0 | 1

4. Secondary Outcome: Pilot Phase + Expansion Phase: Median Progression-free Survival (PFS) (Non-CNS Assessment)
Description: PFS was defined as the time in months from first dose of MM-398 to the date of radiologic disease progression by RECIST per Investigator assessment or death due to any cause, whichever occurred first.
  The date of progression is defined as the earliest date that an overall tumour response of PD or death was recorded. For subjects who did not have a qualifying progressive disease or death, the date of censoring for PFS was the date when the last valid tumour assessment determined a lack of progression. The PFS assessed by the Investigator was analysed using the Kaplan-Meier method, and the median PFS based on non-CNS assessment is presented.
Time Frame: Baseline and every 8 weeks from C1D1 until disease progression, unacceptable toxicity or withdrawal of consent.
Population: The efficacy evaluable population consists of all subjects who received at least 1 dose of MM-398.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pilot Phase: FMX Then MM-398 | Expansion Phase: Cohort 1 | Expansion Phase: Cohort 2 | Expansion Phase: Cohort 3
Number analyzed (Participants) | 13 | 10 | 9 | 10
months | 1.8 [1.0 to 3.6] | 1.9 [1.1 to 15.1] | 4.3 [1.0 to 9.4] | 3.2 [0.9 to 26.1]

5. Secondary Outcome: Expansion Phase: Median PFS for Cohort 3 (CNS Assessment)
Description: PFS was defined as the time in months from first dose of MM-398 to the date of radiologic disease progression by modified RECIST (mRECIST) criteria (CNS disease; Cohort 3) per Investigator assessment or death due to any cause, whichever occurred first.
  The date of progression is defined as the earliest date that an overall tumour response of PD or death was recorded. For subjects who did not have a qualifying progressive disease or death, the date of censoring for PFS was the date when the last valid tumour assessment determined a lack of progression. The PFS assessed by the Investigator was analysed using the Kaplan-Meier method, and the median PFS based on CNS mRECIST assessment is provided for Cohort 3.
Time Frame: Baseline and every 8 weeks from C1D1 until disease progression, unacceptable toxicity or withdrawal of consent.
Population: The efficacy evaluable population consists of all subjects who received at least 1 dose of MM-398. Data is presented for Cohort 3 only which included subjects with brain metastasis, and who underwent CNS assessment using mRECIST criteria.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Expansion Phase: Cohort 3
Number analyzed (Participants) | 10
months | 3.6 [0.9 to 9.6]

6. Secondary Outcome: Pilot Phase + Expansion Phase: BOR (Non-CNS Assessment)
Description: BOR was defined as the best response by RECIST version 1.1 (Non-CNS assessments) criteria per Investigator assessment, recorded from the first dose of MM-398 until disease progression or the start of new anti-cancer therapy and/or surgery.
  Tumour response was classified as CR, PR, SD or PD. Classification of SD required at least 1 assessment of SD at least 4 weeks after starting treatment. Subjects were categorised as not evaluable if there was insufficient data for response classification. The BOR is presented for non-CNS assessments for the Pilot phase and Cohorts 1 - 3.
Time Frame: Baseline and every 8 weeks from C1D1 until disease progression, unacceptable toxicity or withdrawal of consent.
Population: The efficacy evaluable population included all subjects who received at least 1 dose of MM-398.
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Phase: FMX Then MM-398 | Expansion Phase: Cohort 1 | Expansion Phase: Cohort 2 | Expansion Phase: Cohort 3
Number analyzed (Participants) | 13 | 10 | 9 | 10
Participants
  CR | 0 | 0 | 0 | 0
  PR | 1 | 4 | 3 | 3
  SD | 5 | 0 | 3 | 2
  Non-CR/Non-PD | 0 | 0 | 0 | 0
  PD | 5 | 5 | 2 | 3
  Not evaluable | 2 | 1 | 1 | 2

7. Secondary Outcome: Expansion Phase: BOR for Cohort 3 (CNS Assessment)
Description: BOR was defined as the best response by mRECIST criteria (CNS disease; Cohort 3) criteria per Investigator assessment, recorded from the first dose of MM-398 until disease progression or the start of new anti-cancer therapy and/or surgery.
  Tumour response was classified as CR, PR, SD or PD. Classification of SD required at least 1 assessment of SD at least 4 weeks after starting treatment. Subjects were categorised as not evaluable if there was insufficient data for response classification. The BOR is presented for CNS assessments for Cohort 3.
Time Frame: Baseline and every 8 weeks from C1D1 until disease progression, unacceptable toxicity or withdrawal of consent.
Population: The efficacy evaluable population included all subjects who received at least 1 dose of MM-398. Data is presented for Cohort 3 only which included subjects with brain metastasis, and who underwent CNS assessment using mRECIST criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Expansion Phase: Cohort 3
Number analyzed (Participants) | 10
Participants
  CR | 0
  PR | 3
  SD | 3
  Non-CR/Non-PD | 0
  PD | 2
  Not evaluable | 2

8. Secondary Outcome: Pilot Phase + Expansion Phase: Objective Response Rate (ORR) (Non-CNS Assessment)
Description: The ORR was defined as the percentage of subjects with a BOR of either a CR or PR relative to the total number of evaluable subjects. Subjects with insufficient data for response classification were classified as non-responders for objective response. The ORR is presented for non-CNS assessments for the Pilot phase and Cohorts 1 - 3.
Time Frame: Baseline and every 8 weeks from C1D1 until disease progression, unacceptable toxicity or withdrawal of consent.
Population: The efficacy evaluable population included all subjects who received at least 1 dose of MM-398. Percentages are based on the number of subjects in the efficacy evaluable population in the corresponding phase/cohort.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pilot Phase: FMX Then MM-398 | Expansion Phase: Cohort 1 | Expansion Phase: Cohort 2 | Expansion Phase: Cohort 3
Number analyzed (Participants) | 13 | 10 | 9 | 10
percentage of participants | 7.7 [0.19 to 36.03] | 40.0 [12.16 to 73.76] | 33.3 [7.49 to 70.07] | 30.0 [6.67 to 65.25]

9. Secondary Outcome: Expansion Phase: ORR for Cohort 3 (CNS Assessment)
Description: The ORR was defined as the percentage of subjects with a BOR of either a CR or PR relative to the total number of evaluable subjects. Subjects with insufficient data for response classification were classified as non-responders for objective response. The ORR is presented for CNS assessments for Cohort 3.
Time Frame: Baseline and every 8 weeks from C1D1 until disease progression, unacceptable toxicity or withdrawal of consent.
Population: The efficacy evaluable population included all subjects who received at least 1 dose of MM-398. Percentages are based on the number of subjects in the efficacy evaluable population in the corresponding phase/cohort. Data is presented for Cohort 3 which included subjects with brain metastasis, and who underwent CNS assessment using mRECIST criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Expansion Phase: Cohort 3
Number analyzed (Participants) | 10
percentage of participants | 30.0 [6.67 to 65.25]

10. Secondary Outcome: Pilot Phase + Expansion Phase: Median Duration of Objective Response (DOR) (Non-CNS Assessment)
Description: DOR was defined as the time from first documentation of response (CR or PR whichever occurred first, based on Investigator assessment using RECIST criteria) to the date of disease progression or to death due to any cause, whichever occurred first. DOR was computed for subjects who had CR or PR as the BOR. For subjects who did not have a qualifying progressive disease or death, the date of censoring was the date when the last valid tumour assessment determined a lack of progression. The median DOR is presented for non-CNS assessments for the Pilot phase and Cohorts 1-3.
Time Frame: Baseline and every 8 weeks from C1D1 until disease progression, unacceptable toxicity or withdrawal of consent.
Population: The efficacy evaluable population included all subjects who received at least 1 dose of MM-398. Data is presented for the number of subjects who had a BOR classification of CR or PR.
Measure: Median (Full Range); unit: months
Arm/Group | Pilot Phase: FMX Then MM-398 | Expansion Phase: Cohort 1 | Expansion Phase: Cohort 2 | Expansion Phase: Cohort 3
Number analyzed (Participants) | 1 | 4 | 3 | 3
months | 3.84 [3.84 to 3.84] | 7.46 [6.4 to 13.0] | 5.62 [3.7 to 7.4] | 4.14 [0.0 to 22.2]

11. Secondary Outcome: Expansion Phase: Median DOR for Cohort 3 (CNS Assessment)
Description: DOR was defined as the time from first documentation of response (CR or PR whichever occurred first, based on Investigator assessment using mRECIST criteria) to the date of disease progression or to death due to any cause, whichever occurred first. DOR was computed for subjects who had CR or PR as the BOR. For subjects who did not have a qualifying progressive disease or death, the date of censoring was the date when the last valid tumour assessment determined a lack of progression. The median DOR is presented for CNS assessments for Cohort 3.
Time Frame: Baseline and every 8 weeks from C1D1 until disease progression, unacceptable toxicity or withdrawal of consent.
Population: The efficacy evaluable population included all subjects who received at least 1 dose of MM-398. Data is presented for the number of subjects who had a BOR classification of CR or PR. Data is presented for Cohort 3 only which included subjects with brain metastasis, and who underwent CNS assessment using mRECIST criteria.
Measure: Median (Full Range); unit: months
Arm/Group | Expansion Phase: Cohort 3
Number analyzed (Participants) | 3
months | 1.84 [0.0 to 1.9]

12. Secondary Outcome: Pilot Phase + Expansion Phase: Clinical Benefit Response (CBR) (Non-CNS Assessment)
Description: CBR was defined as the percentage of subjects with a BOR characterised as a CR at any time, PR at any time, or SD ≥ 24 weeks relative to the total number of evaluable subjects. The CBR is presented for non-CNS assessments.
Time Frame: Baseline and every 8 weeks from C1D1 until disease progression, unacceptable toxicity or withdrawal of consent.
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pilot Phase: FMX Then MM-398 | Expansion Phase: Cohort 1 | Expansion Phase: Cohort 2 | Expansion Phase: Cohort 3
Number analyzed (Participants) | 13 | 10 | 9 | 10
percentage of participants | 15.4 [1.92 to 45.45] | 40.0 [12.16 to 73.76] | 33.3 [7.49 to 70.07] | 30.0 [6.67 to 65.25]

13. Secondary Outcome: Expansion Phase: CBR for Cohort 3 (CNS Assessment)
Description: CBR was defined as the percentage of subjects with a BOR characterised as a CR at any time, PR at any time, or SD ≥ 24 weeks relative to the total number of evaluable subjects. The CBR is presented for CNS assessment for Cohort 3.
Time Frame: Baseline and every 8 weeks from C1D1 until disease progression, unacceptable toxicity or withdrawal of consent.
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Expansion Phase: Cohort 3
Number analyzed (Participants) | 10
percentage of participants | 50.0 [18.71 to 81.29]

14. Secondary Outcome: Pilot Phase + Expansion Phase: Number of Subjects Who Experienced Treatment Emergent Adverse Events (TEAEs) Related to MM-398
Description: The number of subjects who experienced a TEAE reported to be related to MM-398 by the Investigator are presented for the Pilot and Expansion phases. An AE was considered treatment emergent if it began on or after the first administration of MM-398, started prior to dosing with MM-398 and increased in severity or seriousness after dosing, or started prior to dosing of MM-398 but the causality changed to 'related' after dosing.
Time Frame: From MM-398 treatment start up to 30 days after last dose.
Population: The MM-398 safety population consisted of all subjects who received at least 1 dose of MM-398. Data was combined into 1 arm for the Expansion Phase as all subjects had BC.
Measure: Number; unit: participants
Arm/Group | Pilot Phase: FMX Then MM-398 | Expansion Phase: FMX Then MM-398
Number analyzed (Participants) | 13 | 29
participants | 13 | 28

15. Secondary Outcome: Pilot Phase: Time to Reach Maximum Plasma Concentration of Irinotecan and SN-38 (Tmax)
Description: In Cycle 1 only of the Pilot phase, samples were collected to determine the levels of total irinotecan (liposomal and free drug) and SN-38 (metabolite) in plasma following a dose of 70 mg/m^2 MM-398 FBE (80 mg/m^2 MM-398 salt-base equivalent [SBE]). The pharmacokinetic (PK) analysis was based on non-compartmental analysis. Any plasma concentrations below the lower limit of quantification (LLOQ) were assigned as missing/zero in the data set according to predetermined rules. The LLOQ for irinotecan was 0.140 micrograms per millilitre (mcg/mL), and for SN-38 the LLOQ for the Pilot phase was 0.441 nanograms per millilitre (ng/mL). The median tmax is presented for the Pilot phase.
Time Frame: Pilot phase: C1D1 pre-MM-398 infusion, end of infusion, post-infusion (2, 72, 168 hours); C1D15 pre-infusion; 30 days follow-up visit.
Population: The PK set included subjects who received at least 1 dose of MM-398, blood samples were collected at the predefined points (with no major protocol deviations affecting PK variables & sufficient number of plasma concentrations to estimate main PK parameters [Cmax, AUC]); analysis was within the sample stability period to estimate main PK parameters.
Measure: Median (Full Range); unit: hours
Arm/Group | Pilot Phase: FMX Then MM-398
Number analyzed (Participants) | 13
hours
  Irinotecan | 1.72 [1.52 to 3.20]
  SN-38 | 3.20 [1.65 to 75.22]

16. Secondary Outcome: Expansion Phase: Irinotecan and SN-38 Tmax
Description: For the Expansion phase, samples were collected to determine the levels of total irinotecan (liposomal and free drug) and SN-38 (metabolite) in plasma and data is presented for Cycles 1 to 3 by dose received for each cycle (depending on dose titration): 35 to 70 mg/m^2 MM-398 FBE (40 to 80 mg/m^2 MM-398 SBE). The PK analysis was based on non-compartmental analysis. Any plasma concentrations below the LLOQ were assigned as missing/zero in the data set according to predetermined rules. The LLOQ for irinotecan was 0.140 mcg/mL and for SN-38 the LLOQ for the Expansion phase was 0.600 ng/mL. The median tmax is presented for dose levels in the Expansion phase for which data was collected. PK results for subjects in all cohorts of the Expansion Phase were combined for those on the same cycle and at the same dose. The total number of subjects evaluated in the PK set for the Expansion Phase was 21, with different numbers evaluated for each cycle/dose.
Time Frame: Expansion phase: Cycles 1-3 pre-MM-398 infusion, end of infusion, post-infusion (2, 48,168 hours); D15 pre-infusion; 30 days follow-up visit.
Population: as for outcome 15
Measure: Median (Full Range); unit: hours
Arm/Group | Expansion Phase: FMX Then MM-398
Number analyzed (Participants) | 21
hours
  Irinotecan: Cycle 1 40 mg/m^2 SBE: number analyzed (Participants) | 1
  Irinotecan: Cycle 1 40 mg/m^2 SBE | NA [3.88 to 3.88] — Descriptive statistics could not be determined for this sample size and therefore the median value was not calculated.
  Irinotecan: Cycle 1 60 mg/m^2 SBE: number analyzed (Participants) | 12
  Irinotecan: Cycle 1 60 mg/m^2 SBE | 1.71 [1.52 to 3.67]
  Irinotecan: Cycle 1 80 mg/m^2 SBE: number analyzed (Participants) | 5
  Irinotecan: Cycle 1 80 mg/m^2 SBE | 1.73 [1.63 to 1.80]
  Irinotecan: Cycle 2 40 mg/m^2 SBE: number analyzed (Participants) | 1
  Irinotecan: Cycle 2 40 mg/m^2 SBE | NA [1.98 to 1.98] — Descriptive statistics could not be determined for this sample size and therefore the median value was not calculated.
  Irinotecan: Cycle 2 60 mg/m^2 SBE: number analyzed (Participants) | 12
  Irinotecan: Cycle 2 60 mg/m^2 SBE | 3.03 [1.58 to 3.62]
  Irinotecan: Cycle 2 80 mg/m^2 SBE: number analyzed (Participants) | 5
  Irinotecan: Cycle 2 80 mg/m^2 SBE | 2.12 [1.70 to 3.55]
  Irinotecan: Cycle 3 40 mg/m^2 SBE: number analyzed (Participants) | 2
  Irinotecan: Cycle 3 40 mg/m^2 SBE | NA [1.68 to 2.50] — Descriptive statistics could not be determined for this sample size and therefore the median value was not calculated.
  Irinotecan: Cycle 3 60 mg/m^2 SBE: number analyzed (Participants) | 8
  Irinotecan: Cycle 3 60 mg/m^2 SBE | 3.26 [1.63 to 48.33]
  Irinotecan: Cycle 3 80 mg/m^2 SBE: number analyzed (Participants) | 4
  Irinotecan: Cycle 3 80 mg/m^2 SBE | 2.47 [1.50 to 6.92]
  SN-38: Cycle 1 60 mg/m^2 SBE: number analyzed (Participants) | 6
  SN-38: Cycle 1 60 mg/m^2 SBE | 3.08 [1.57 to 40.82]
  SN-38: Cycle 2 60 mg/m^2 SBE: number analyzed (Participants) | 4
  SN-38: Cycle 2 60 mg/m^2 SBE | 25.88 [3.08 to 67.42]
  SN-38: Cycle 2 80 mg/m^2 SBE: number analyzed (Participants) | 1
  SN-38: Cycle 2 80 mg/m^2 SBE | NA [1.70 to 1.70] — Descriptive statistics could not be determined for this sample size and therefore the median value was not calculated.
  SN-38: Cycle 3 60 mg/m^2 SBE: number analyzed (Participants) | 4
  SN-38: Cycle 3 60 mg/m^2 SBE | 31.29 [1.65 to 44.95]
  SN-38: Cycle 3 80 mg/m^2 SBE: number analyzed (Participants) | 1
  SN-38: Cycle 3 80 mg/m^2 SBE | NA [3.27 to 3.27] — Descriptive statistics could not be determined for this sample size and therefore the median value was not calculated.

17. Secondary Outcome: Pilot Phase: Maximum Observed Plasma Concentration of Irinotecan (Cmax)
Description: In Cycle 1 only of the Pilot phase, samples were collected to determine the levels of total irinotecan (liposomal and free drug) in plasma following a dose of 70 mg/m^2 MM-398 FBE (80 mg/m^2 MM-398 SBE). The PK analysis was based on non-compartmental analysis. Any plasma concentrations below the LLOQ were assigned as missing/zero in the data set according to predetermined rules. The LLOQ for irinotecan was 0.140 mcg/mL. The mean Cmax is presented for the Pilot phase.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Mean (Full Range); unit: mcg/mL
Arm/Group | Pilot Phase: FMX Then MM-398
Number analyzed (Participants) | 13
mcg/mL | 39.0 [20.4 to 47.1]

18. Secondary Outcome: Pilot Phase: SN-38 Cmax
Description: In Cycle 1 only of the Pilot phase, samples were collected to determine the levels of SN-38 (metabolite) in plasma following a dose of 70 mg/m^2 MM-398 FBE (80 mg/m^2 MM-398 SBE). The PK analysis was based on non-compartmental analysis. Any plasma concentrations below the LLOQ were assigned as missing/zero in the data set according to predetermined rules. The LLOQ for SN-38 for the Pilot phase was 0.441 ng/mL. The mean Cmax is presented for the Pilot phase.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Pilot Phase: FMX Then MM-398
Number analyzed (Participants) | 13
ng/mL | 2.40 [1.52 to 3.62]

19. Secondary Outcome: Expansion Phase: Irinotecan Cmax
Description: For the Expansion phase, samples were collected to determine the levels of total irinotecan (liposomal and free drug) in plasma and data is presented for Cycles 1 to 3 by dose received for each cycle (depending on dose titration): 35 to 70 mg/m^2 MM-398 FBE (40 to 80 mg/m^2 MM-398 SBE). The PK analysis was based on non-compartmental analysis. Any plasma concentrations below the LLOQ were assigned as missing/zero in the data set according to predetermined rules. The LLOQ for irinotecan was 0.140 mcg/mL. The mean Cmax is presented for the Expansion phase. PK results for subjects in all cohorts of the Expansion Phase were combined for those on the same cycle and at the same dose. The total number of subjects evaluated in the PK set for the Expansion Phase was 21, with different numbers evaluated for each cycle/dose.
Time Frame: as for outcome 16
Population: as for outcome 15
Measure: Mean (Full Range); unit: mcg/mL
Arm/Group | Expansion Phase: FMX Then MM-398
Number analyzed (Participants) | 21
mcg/mL
  Cycle 1 40 mg/m^2 SBE: number analyzed (Participants) | 1
  Cycle 1 40 mg/m^2 SBE | NA [21.7 to 21.7] — Descriptive statistics could not be determined for this sample size and therefore the mean value was not calculated.
  Cycle 1 60 mg/m^2 SBE: number analyzed (Participants) | 12
  Cycle 1 60 mg/m^2 SBE | 28.1 [20.8 to 40.4]
  Cycle 1 80 mg/m^2 SBE: number analyzed (Participants) | 5
  Cycle 1 80 mg/m^2 SBE | 44.4 [34.2 to 56.4]
  Cycle 2 40 mg/m^2 SBE: number analyzed (Participants) | 1
  Cycle 2 40 mg/m^2 SBE | NA [22.1 to 22.1] — Descriptive statistics could not be determined for this sample size and therefore the mean value was not calculated.
  Cycle 2 60 mg/m^2 SBE: number analyzed (Participants) | 12
  Cycle 2 60 mg/m^2 SBE | 30.4 [15.7 to 37.3]
  Cycle 2 80 mg/m^2 SBE: number analyzed (Participants) | 5
  Cycle 2 80 mg/m^2 SBE | 46.6 [34.2 to 55.8]
  Cycle 3 40 mg/m^2 SBE: number analyzed (Participants) | 2
  Cycle 3 40 mg/m^2 SBE | NA [18.3 to 19.9] — Descriptive statistics could not be determined for this sample size and therefore the mean value was not calculated.
  Cycle 3 60 mg/m^2 SBE: number analyzed (Participants) | 8
  Cycle 3 60 mg/m^2 SBE | 30.3 [17.5 to 40.8]
  Cycle 3 80 mg/m^2 SBE: number analyzed (Participants) | 4
  Cycle 3 80 mg/m^2 SBE | 45.8 [38.6 to 51.5]

20. Secondary Outcome: Expansion Phase: SN-38 Cmax
Description: For the Expansion phase, samples were collected to determine the levels of SN-38 (metabolite) in plasma and data is presented for Cycles 1 to 3 by dose received for each cycle (depending on dose titration): 35 to 70 mg/m^2 MM-398 FBE (40 to 80 mg/m^2 MM-398 SBE). The PK analysis was based on non-compartmental analysis. Any plasma concentrations below the LLOQ were assigned as missing/zero in the data set according to predetermined rules. The LLOQ for SN-38 for the Expansion phase was 0.600 ng/mL. The mean Cmax is presented for dose levels in the Expansion phase for which data was collected. PK results for subjects in all cohorts of the Expansion Phase were combined for those on the same cycle and at the same dose. The total number of subjects evaluated in the PK set for the Expansion Phase was 21, with different numbers evaluated for each cycle/dose.
Time Frame: as for outcome 16
Population: as for outcome 15
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Expansion Phase: FMX Then MM-398
Number analyzed (Participants) | 21
ng/mL
  Cycle 1 60 mg/m^2 SBE: number analyzed (Participants) | 6
  Cycle 1 60 mg/m^2 SBE | 3.08 [2.01 to 5.23]
  Cycle 2 60 mg/m^2 SBE: number analyzed (Participants) | 4
  Cycle 2 60 mg/m^2 SBE | 3.63 [1.74 to 7.62]
  Cycle 2 80 mg/m^2 SBE: number analyzed (Participants) | 1
  Cycle 2 80 mg/m^2 SBE | NA [4.14 to 4.14] — Descriptive statistics could not be determined for this sample size and therefore the mean value was not calculated.
  Cycle 3 60 mg/m^2 SBE: number analyzed (Participants) | 4
  Cycle 3 60 mg/m^2 SBE | 2.60 [1.03 to 3.55]
  Cycle 3 80 mg/m^2 SBE: number analyzed (Participants) | 1
  Cycle 3 80 mg/m^2 SBE | NA [3.08 to 3.08] — Descriptive statistics could not be determined for this sample size and therefore the mean value was not calculated.

21. Secondary Outcome: Pilot Phase: Area Under the Plasma Concentration Time Curve From Time Zero to Last Quantifiable Concentration (AUC[0-tlast]) for Irinotecan
Description: In Cycle 1 only of the Pilot phase, samples were collected to determine the levels of total irinotecan (liposomal and free drug) in plasma following a dose of 70 mg/m^2 MM-398 FBE (80 mg/m^2 MM-398 SBE). The PK analysis was based on non-compartmental analysis. Any plasma concentrations below the LLOQ were assigned as missing/zero in the data set according to predetermined rules. The LLOQ for irinotecan was 0.140 mcg/mL. The mean AUC(0-tlast) is presented for the Pilot phase.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Mean (Full Range); unit: mcg*hours/mL (mcg*h/mL)
Arm/Group | Pilot Phase: FMX Then MM-398
Number analyzed (Participants) | 13
mcg*hours/mL (mcg*h/mL) | 1721 [293 to 3758]

22. Secondary Outcome: Pilot Phase: SN-38 AUC(0-tlast)
Description: In Cycle 1 only of the Pilot phase, samples were collected to determine the levels of SN-38 (metabolite) in plasma following a dose of 70 mg/m^2 MM-398 FBE (80 mg/m^2 MM-398 SBE). The PK analysis was based on non-compartmental analysis. Any plasma concentrations below the LLOQ were assigned as missing/zero in the data set according to predetermined rules. The LLOQ for SN-38 for the Pilot phase was 0.441 ng/mL. The mean AUC(0-tlast) is presented for the Pilot phase.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Mean (Full Range); unit: ng*h/mL
Arm/Group | Pilot Phase: FMX Then MM-398
Number analyzed (Participants) | 13
ng*h/mL | 212 [89.1 to 380]

23. Secondary Outcome: Expansion Phase: Irinotecan AUC(0-tlast)
Description: For the Expansion phase, samples were collected to determine the levels of total irinotecan (liposomal and free drug) in plasma and data is presented for Cycles 1 to 3 by dose received for each cycle (depending on dose titration): 35 to 70 mg/m^2 MM-398 FBE (40 to 80 mg/m^2 MM-398 SBE). The PK analysis was based on non-compartmental analysis. Any plasma concentrations below the LLOQ were assigned as missing/zero in the data set according to predetermined rules. The LLOQ for irinotecan was 0.140 mcg/mL. The mean AUC(0-tlast) is presented for the Expansion phase. PK results for subjects in all cohorts of the Expansion Phase were combined for those on the same cycle and at the same dose. The total number of subjects evaluated in the PK set for the Expansion Phase was 21, with different numbers evaluated for each cycle/dose.
Time Frame: as for outcome 16
Population: as for outcome 15
Measure: Mean (Full Range); unit: mcg*h/mL
Arm/Group | Expansion Phase: FMX Then MM-398
Number analyzed (Participants) | 21
mcg*h/mL
  Cycle 1 40 mg/m^2 SBE: number analyzed (Participants) | 1
  Cycle 1 40 mg/m^2 SBE | NA [976 to 976] — Descriptive statistics could not be determined for this sample size and therefore the mean value was not calculated.
  Cycle 1 60 mg/m^2 SBE: number analyzed (Participants) | 12
  Cycle 1 60 mg/m^2 SBE | 1430 [230 to 3301]
  Cycle 1 80 mg/m^2 SBE: number analyzed (Participants) | 4
  Cycle 1 80 mg/m^2 SBE | 1530 [541 to 2273]
  Cycle 2 40 mg/m^2 SBE: number analyzed (Participants) | 1
  Cycle 2 40 mg/m^2 SBE | NA [1185 to 1185] — Descriptive statistics could not be determined for this sample size and therefore the mean value was not calculated.
  Cycle 2 60 mg/m^2 SBE: number analyzed (Participants) | 12
  Cycle 2 60 mg/m^2 SBE | 1589 [204 to 2963]
  Cycle 2 80 mg/m^2 SBE: number analyzed (Participants) | 4
  Cycle 2 80 mg/m^2 SBE | 1788 [902 to 2266]
  Cycle 3 40 mg/m^2 SBE: number analyzed (Participants) | 2
  Cycle 3 40 mg/m^2 SBE | NA [426 to 969] — Descriptive statistics could not be determined for this sample size and therefore the mean value was not calculated.
  Cycle 3 60 mg/m^2 SBE: number analyzed (Participants) | 6
  Cycle 3 60 mg/m^2 SBE | 1700 [325 to 3001]
  Cycle 3 80 mg/m^2 SBE: number analyzed (Participants) | 2
  Cycle 3 80 mg/m^2 SBE | NA [1345 to 2288] — Descriptive statistics could not be determined for this sample size and therefore the mean value was not calculated.

24. Secondary Outcome: Expansion Phase: SN-38 AUC(0-tlast)
Description: For the Expansion phase, samples were collected to determine the levels of SN-38 (metabolite) in plasma and data is presented for Cycles 1 to 3 by dose received for each cycle (depending on dose titration): 35 to 70 mg/m^2 MM-398 FBE (40 to 80 mg/m^2 MM-398 SBE). The PK analysis was based on non-compartmental analysis. Any plasma concentrations below the LLOQ were assigned as missing/zero in the data set according to predetermined rules. The LLOQ for SN-38 for the Expansion phase was 0.600 ng/mL. The mean AUC(0-tlast) is presented for dose levels in the Expansion phase for which data was collected. PK results for subjects in all cohorts of the Expansion Phase were combined for those on the same cycle and at the same dose. The total number of subjects evaluated in the PK set for the Expansion Phase was 21, with different numbers evaluated for each cycle/dose.
Time Frame: as for outcome 16
Population: as for outcome 15
Measure: Mean (Full Range); unit: ng*h/mL
Arm/Group | Expansion Phase: FMX Then MM-398
Number analyzed (Participants) | 21
ng*h/mL
  Cycle 1 60 mg/m^2 SBE: number analyzed (Participants) | 5
  Cycle 1 60 mg/m^2 SBE | 237 [40.5 to 599]
  Cycle 2 60 mg/m^2 SBE: number analyzed (Participants) | 2
  Cycle 2 60 mg/m^2 SBE | NA [237 to 353] — Descriptive statistics could not be determined for this sample size and therefore the mean value was not calculated.
  Cycle 2 80 mg/m^2 SBE: number analyzed (Participants) | 1
  Cycle 2 80 mg/m^2 SBE | NA [354 to 354] — Descriptive statistics could not be determined for this sample size and therefore the mean value was not calculated.
  Cycle 3 60 mg/m^2 SBE: number analyzed (Participants) | 3
  Cycle 3 60 mg/m^2 SBE | 214 [146 to 295]
  Cycle 3 80 mg/m^2 SBE: number analyzed (Participants) | 1
  Cycle 3 80 mg/m^2 SBE | NA [119 to 119] — Descriptive statistics could not be determined for this sample size and therefore the mean value was not calculated.

ADVERSE EVENTS:
Time Frame: TEAEs were collected from MM-398 treatment start to end of study (approximately 6 years). An AE was considered treatment emergent if it began on or after the first administration of MM-398, started prior to dosing with MM-398 and increased in severity or seriousness after dosing, or started prior to dosing of MM-398 but the causality changed to 'related' after dosing.
Description: TEAEs are presented for the MM-398 safety population which included all subjects who received at least 1 dose of MM-398. All analyses using this population were based on the treatment actually received. All cause mortality is presented for the safety population which included all subjects who received at least 1 dose of FMX or MM-398, and the subjects affected received FMX only. Data was combined into 1 arm for the Expansion Phase as all subjects had BC.
Arm/Group | Pilot Phase: FMX Then MM-398 | Expansion Phase: FMX Then MM-398
All-Cause Mortality (participants affected / at risk) | 2/15 | 1/30
Serious Adverse Events (participants affected / at risk) | 4/13 | 17/29
Other Adverse Events (participants affected / at risk) | 13/13 | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pilot Phase: FMX Then MM-398 (N=13) | Expansion Phase: FMX Then MM-398 (N=29)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 5 (5)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (4)
Coccidioidomycosis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 3 (3)
Fatigue (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pilot Phase: FMX Then MM-398 (N=13) | Expansion Phase: FMX Then MM-398 (N=29)
Diarrhoea (Gastrointestinal disorders) | 9 | 25
Nausea (Gastrointestinal disorders) | 9 | 15
Vomiting (Gastrointestinal disorders) | 7 | 11
Constipation (Gastrointestinal disorders) | 5 | 5
Abdominal pain (Gastrointestinal disorders) | 2 | 6
Dyspepsia (Gastrointestinal disorders) | 2 | 2
Flatulence (Gastrointestinal disorders) | 1 | 3
Stomatitis (Gastrointestinal disorders) | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 2
Oral pain (Gastrointestinal disorders) | 0 | 3
Ascites (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 11
Decreased appetite (Metabolism and nutrition disorders) | 3 | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 6
Dehydration (Metabolism and nutrition disorders) | 2 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 2
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0
Fatigue (General disorders) | 3 | 17
Asthenia (General disorders) | 0 | 3
Oedema peripheral (General disorders) | 1 | 3
Chills (General disorders) | 1 | 1
Mucosal inflammation (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Headache (Nervous system disorders) | 3 | 6
Dizziness (Nervous system disorders) | 2 | 2
Dysgeusia (Nervous system disorders) | 2 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 3
Urinary tract infection (Infections and infestations) | 3 | 4
Pneumonia (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Enterocolitis infection (Infections and infestations) | 1 | 0
Lymphangitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Skin candida (Infections and infestations) | 1 | 0
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 6
Neutrophil count decreased (Investigations) | 0 | 5
Aspartate aminotransferase increased (Investigations) | 0 | 4
Weight decreased (Investigations) | 0 | 4
Blood alkaline phosphatase increased (Investigations) | 0 | 3
White blood cell count decreased (Investigations) | 0 | 3
Lymphocyte count decreased (Investigations) | 0 | 3
Blood phosphorous decreased (Investigations) | 0 | 2
Transaminases increased (Investigations) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 5 | 7
Neutropenia (Blood and lymphatic system disorders) | 4 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 6
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 4
Insomnia (Psychiatric disorders) | 0 | 3
Depression (Psychiatric disorders) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 2
Blepharospasm (Eye disorders) | 0 | 2
Vision blurred (Eye disorders) | 0 | 2
Hypotension (Vascular disorders) | 0 | 3
Hypertension (Vascular disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
Data for the subjects in the 3 Expansion Phase cohorts were combined when presenting results for the overall Expansion Phase because all cohorts were defined in the protocol to contain subjects with BC.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-02-28): https://cdn.clinicaltrials.gov/large-docs/53/NCT01770353/SAP_000.pdf
  • Study Protocol (2017-04-03): https://cdn.clinicaltrials.gov/large-docs/53/NCT01770353/Prot_001.pdf